CLINICAL TRIAL: NCT06447805
Title: "A Pilot Study Assessing Feasibility of a Randomized Trial Comparing the Effect of Early Double Sequential Defibrillation as Soon as Possible in OHCA With a Shockable Rhythm (VT/VF) Compared to Standard Defibrillation"
Brief Title: Early Double Sequential Defibrillation in Out-of-hospital Cardiac Arrest
Acronym: DOUBLE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Riva, Principal Investigator, M.D., Ph.D. Center for resuscitation Scinence, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIV-ID-24-01-045759
Record Dates: First submitted 2024-05-29; First posted 2024-06-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrest; Fibrillation, Ventricular; Sudden Cardiac Death; Sudden Cardiac Arrest
Keywords: Cardiopulmonary resuscitation; Defibrillation; Double sequential defibrillation
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation; Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: Academic, investigator initiated, open-label pilot study with a randomized controlled trial (RCT) design and 3:1 allocation (3 intervention: 1 standard).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double Sequential Defibrillation (DSD) (Experimental): If the patient is randomized to the DSD group, the ambulance crew team will apply the second defibrillator with electrodes placed in the A-P position as soon as possible.
  Defibrillation is performed by one person defibrillating both defibrillators in a sequential manner "Double Sequential Defibrillation" (DSD). All consecutive defibrillations will thereafter be performed with the DSD strategy until ROSC, termination of resuscitation or decision to move the patient to hospital.
  Interventions: Device: Double Sequential Defibrillation (DSD)
- Standard defibrillation (Active Comparator): If the patient is randomized to the standard defibrillation group, the ambulance crew team will continue Advanced life support in accordance with standard of care and continue to perform standard defibibrillation using one defibrillator. All consecutive defibrillations will thereafter be performed with the standard defibrillation strategy until ROSC, termination of resuscitation or decision to move the patient to hospital.
  Interventions: Device: Standard defibrillation

INTERVENTIONS:
Device: Double Sequential Defibrillation (DSD) — The second defibrillator will be applyed with electrodes placed in the A-P position
  Arms: Double Sequential Defibrillation (DSD)
Device: Standard defibrillation — Standard defibrillation uning one defibrillator
  Arms: Standard defibrillation

SUMMARY:
Some of the patients affected by Out-of-hospital cardiac arrest (OHCA) with ventricular fibrillation (VF)/ventricular tachycardia (VT) do not respond to initial defibrillation. The survival decreases with number of defibrillations required to terminate VF/VT. In 2022, one prospective cluster randomized trial showed increased survival among (OHCA) patients in refractory VF using Double Sequential Defibrillation (DSD).

To evaluate feasibility and safety this randomized pilot trial will compare the effect of double defibrillation strategy initiated as soon as possible after the first defibrillation with continued resuscitation using standard defibrillation, in patients with Out of Hospital Cardiac arrest (OHCA). The results from this pilot trial will form the basis for design of a larger multicenter survival study.

DETAILED DESCRIPTION:
The Dubbel-D study is an academic, investigator initiated, open-label pilot study with a randomized controlled trial (RCT) design conducted in the prehospital emergency medical services, i.e. ambulance organizations. The trial will be conducted by participating ambulance units attending OHCA´s. These units will perform screening for inclusion, randomization, intervention or control treatment and initial follow-up.

In all cases of OHCA a defibrillator should always be attached with the standard pad placement, anterio-lateral (A-L) position first. This is in accordance with standard of care. If there is VT/VF or an automated external defibrillator (AED) suggests defibrillation, defibrillation should be performed, and immediate chest compressions resumed. Thereafter, the patient can be screened for inclusion. If two study specific defibrillators (Corpulse 3) on site and no exclusion criteria (age below 18 years, obvious pregnancy, known preexisting Do Not Attempt Resuscitation order) the patient can be included and randomized.

Randomization will be performed by drawing a scratch-card with concealed allocation that will be stored with the EMS defibrillators. All scratch-cards will be pre-randomized in a 3:1 ratio in blocks consisting of 4-8-12 and stratified by region and ambulance provider.

If the patient is randomized to the intervention group, the ambulance crew team will apply the second defibrillator with electrodes placed in the anterio-posterior (A-P) position as soon as possible. Defibrillation is performed by one person defibrillating both defibrillators in a sequential manner "Double Sequential Defibrillation" (DSD). All consecutive defibrillations will thereafter be performed with the DSD strategy until ROSC, termination of resuscitation or decision to move the patient to hospital.

If randomized to the control group, the ambulance crew team will continue Advanced Life Support (ACLS) in accordance with standard of care. Defibrillation is performed with standard electrode placement (A-L position) using a single defibrillator. If an AED is the first defibrillator attached to the patient, the ambulance crew should shift from an AED to their own manual defibrillator, but the mode of defibrillation should remain in A-L position and only one defibrillator should be used for each defibrillation and continue until ROSC, termination of resuscitation or decision to move the patient to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-Hospital patients with Ventricular Fibrillation/ Ventricular Tachycardia at rhythm analysis after ambulance arrival and at least one defibrillation performed in standard (Antero-Lateral) position

Exclusion Criteria:

* Age below 18 years
* Obvious pregnancy
* Known preexisting Do Not Attempt Resuscitation order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of early double sequential external defibrillation (DSD) | day 1
  Number of EMS defibrillations prior to randomization (target > 80% before third defibrillation)
Adherence to double sequential external defibrillation (DSD) | day 1
  Among patients randomized to DSD, proportion that received DSD (target > 80%)
Cross-over | day 1
  Among patients randomized to standard, proportion that received DSD (target < 10%)
Feasibility of double sequential external defibrillation (DSD) | day 1
  Proportion of eligible patients included and randomized (target > 80%)
Safety of double sequential external defibrillation | day 1
  Major adverse events (e.g. defibrillator malfunction)
Safety of CPR during double sequential external defibrillation | day 1
  Chest compression fraction (hands off time during CPR, target > 80% in both groups)

SECONDARY OUTCOMES:
Return of spontaneous circulation (ROSC) | day 1
  Proportion of patients with sustained return of spontaneous circulation (ROSC) at hospital arrival
Number of defibrillations to sustained ROSC | day 1
  Total number of defibrillations to sustained ROSC
Survival to hospital admission | day 1
  Pateint is admitted to hospital alive
Survival to discharge | day 1-180
  Survival to hospital discharge
30 day survival | day 30
  Survival at 30 days
Neurological function at 30 days | day 30
  Neurological function (modified Rankin Scale, mRS 1-6, and Cerebral Performance Category, CPC 1-5) at 30 days
Neurological function and Health related Quality of life at 90 and 180 days | day 90 and 180
  Neurological function (modifiied Rankin Scale and Cerebral Performance Category) and Health-related Quality of life at 90 and 180 days (CPC 1-5, mRS 1-6)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Riva, MD, PhD, Principal Investigator — Karolinska Institutet; Akil Awad, MD, PhD, Principal Investigator — Karolinska Institutet; Andreas Claesson, RN, PhD, Study Chair — Karolinska Institutet; Carl Magnusson, RN, PhD, Study Chair — Sahlgrenska University; Leif Svensson, MD, PhD, Study Chair — Karolinska Institutet; Johan Israelsson, RN, PhD, Study Chair — Linné University; Emma Blick-Nordqvist, MD, Study Chair — Karolinska Institutet; Martin Jonsson, Msc, PhD, Study Chair — Karolinska Institutet; Jacob Hollenberg, MD, PhD, Study Chair — Karolinska Institutet; Sheldon Cheskes, MD, Study Chair — University of Toronto
Locations (3):
- Sweden (3):
  - Emergency medical services Region Halland, Halmstad, Halland County
  - Sahlgrenska Universitetssjukhuset, Ambulans och Prehospital Akutsjukvård, Gothenburg, Västra Götalandsregionen
  - Sjukhusen i väster, ambulanssjukvården Alingsås/Lerum, Alingsås, Västra Götalandsregionen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheskes S, Verbeek PR, Drennan IR, McLeod SL, Turner L, Pinto R, Feldman M, Davis M, Vaillancourt C, Morrison LJ, Dorian P, Scales DC. Defibrillation Strategies for Refractory Ventricular Fibrillation. N Engl J Med. 2022 Nov 24;387(21):1947-1956. doi: 10.1056/NEJMoa2207304. Epub 2022 Nov 6. PMID 36342151

DOCUMENTS (1):
  • Study Protocol (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT06447805/Prot_001.pdf